CLINICAL TRIAL: NCT03225105
Title: A Phase I, Open-label, Uncontrolled, Multicenter, Dose-escalation Study of M3541 in Combination With Palliative Radiotherapy in Subjects With Solid Tumors
Brief Title: M3541 in Combination With Radiotherapy in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early per sponsor decision to halt further development of M3541 due to pharmaceutical and PK/pharmacodynamics properties that precluded further clinical development.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200770_0001
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; M3541; Palliative radiotherapy; Adenosine triphosphate-competitive inhibitor

STUDY DESIGN:
Intervention Model Description: Subsequent cohorts of patients treated at different dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- M3541 50 mg + RT (Experimental): Participants received 50 milligrams (mg) M3541 orally once per fraction day (FD) in combination with palliative radiotherapy (RT) administered in fraction of 30 Gray (Gy) given in 10 fractions of 3 Gy/FD on FD 1 to FD 10, for 2 consecutive calendar weeks (ie, Monday through Friday, with the intervening Saturday and Sunday as M3541 / RT holidays).
  Interventions: Drug: M3541; Radiation: Palliative Radiotherapy (RT)
- M3541 100 mg + RT (Experimental): Participants received 100 mg M3541 orally once per FD in combination with palliative RT administered in fraction of 30 Gray (Gy) given in 10 fractions of 3 Gy/FD on FD 1 to FD 10 for 2 consecutive calendar weeks (ie, Monday through Friday, with the intervening Saturday and Sunday as M3541 / RT holidays).
  Interventions: Drug: M3541; Radiation: Palliative Radiotherapy (RT)
- M3541 200 mg + RT (Experimental): Participants received 200 mg M3541 orally once per FD in combination with palliative RT administered in fraction of 30 Gray (Gy) given in 10 fractions of 3 Gy/FD on FD 1 to FD 10 for 2 consecutive calendar weeks (ie, Monday through Friday, with the intervening Saturday and Sunday as M3541 / RT holidays).
  Interventions: Drug: M3541; Radiation: Palliative Radiotherapy (RT)
- M3541 300 mg + RT (Experimental): Participants received 300 mg M3541 orally once per FD in combination with palliative RT administered in fraction of 30 Gray (Gy) given in 10 fractions of 3 Gy/FD on FD 1 to FD 10 for 2 consecutive calendar weeks (ie, Monday through Friday, with the intervening Saturday and Sunday as M3541 / RT holidays).
  Interventions: Drug: M3541; Radiation: Palliative Radiotherapy (RT)

INTERVENTIONS:
Drug: M3541 — Participants received M3541 orally once per fraction day (FD) for two consecutive calendar weeks (that is, Monday through Friday, with Saturday and Sunday as M3541 holidays).
Radiation: Palliative Radiotherapy (RT) — Participants received RT dose of 30 Gray (Gy) given in 10 fractions (3 Gy given per fraction day) administered over two consecutive calendar weeks (that is, Monday through Friday, with Saturday and Sunday as RT holidays).

SUMMARY:
This dose-escalation study evaluated the safety, tolerability, pharmacokinetic (PK), pharmacodynamic, and explore antitumor activity of M3541 in combination with fractionated palliative radiotherapy (RT) in participants with solid tumors with malignant lesions in the thorax, abdominal cavity, head and neck region, or extremities likely to benefit from palliative RT.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have solid tumors with malignant lesions in the thorax, abdominal cavity, head and neck region, or extremities (any histology) likely to benefit from palliative radiotherapy; participants requiring palliative RT for lesions in the spine or lesions adjacent to the spinal cord are excluded from this study
* Eastern Cooperative Oncology Group performance status (ECOG PS) =< 2
* Life expectancy >= 3 months
* Adequate hematologic, hepatic, and renal function
* Agree to use highly effective contraception (that is, methods with a failure rate of less than 1 percent per year) if the participant is male or a female of childbearing potential (female partners of childbearing potential of male participants must also agree to use highly effective contraception)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Use of other anticancer therapy within 15 days before the first dose of M3541 administration and should not be within the "at risk follow-up period" for that specific anticancer therapy. The use of any investigational agent is not allowed within 28 days before the first dose of M3541
* Residual toxicity due to previous anticancer therapy with no return to baseline or =< Grade 1 (except alopecia) according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03
* Extensive prior RT on more than 30 percent of bone marrow reserves (by Investigator judgment), or prior bone marrow/stem cell transplantation within 5 years before study start
* Prior RT to the same region that would be irradiated in this study
* Participants at increased risk for radiation toxicities, such as known collagen vascular disease (example, scleroderma, Sjogren's disease, etc) or other inherited radiation hypersensitivity syndromes (example, Gorlin syndrome, Fanconi anemia, ataxia-telangiectasia, etc.)
* Surgical intervention within 28 days prior to the first dose of M3541 administration
* Known central nervous system metastases causing clinical symptoms or metastases that require therapeutic intervention. Participants with a history of treated central nervous system (CNS) metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy. Participants with CNS metastases incidentally detected during Screening that do not cause clinical symptoms and for which standard of care suggests no therapeutic intervention is indicated, should be discussed with the Sponsor Medical Responsible
* Active difficulty swallowing, malabsorption or other chronic gastrointestinal disease or conditions (including pancreas deficiency requiring Creon therapy) that may hamper compliance and/or absorption of M3541
* Participants currently receiving or unable to stop using medications or herbal supplements known to be potent inhibitors of cytochrome P450 (CYP) 3A and / or P-glycoprotein (P-gp) (CYP and / P-gp must stop at least 1 week before treatment with M3541) or potent inducers of CYP3A or P-gp (must stop at least 3 weeks before treatment with M3541) or drugs mainly metabolized by CYP3A with a narrow therapeutic index (must stop at least 1 day prior).
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (5):
- United States (5):
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Waqar SN, Robinson C, Olszanski AJ, Spira A, Hackmaster M, Lucas L, Sponton L, Jin H, Hering U, Cronier D, Grinberg M, Seithel-Keuth A, Diaz-Padilla I, Berlin J. Phase I trial of ATM inhibitor M3541 in combination with palliative radiotherapy in patients with solid tumors. Invest New Drugs. 2022 Jun;40(3):596-605. doi: 10.1007/s10637-022-01216-8. Epub 2022 Feb 12. PMID 35150356
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200770_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This dose-escalation study was planned to be conducted as per 3 dosing schedules for M3541 including M3541 once per Fraction Day daily, M3541 twice and thrice weekly in combination with fractionated RT given in 10 fractions. However, due to early termination of the study, 2 intermittent schedules (thrice weekly and twice weekly) were never opened and did not enroll any participants.
Period: Overall Study
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Started | 3 | 4 | 5 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Death | 0 | 4 | 2 | 0
Not completed — Study termination per Sponsor Decision | 2 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Groups:
- Total: Total of all reporting groups
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT | Total
Number analyzed (Participants) | 3 | 4 | 5 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (3.8) | 67 (6.3) | 66 (7.4) | 47 (10.1) | 62 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 2 | 8
  Male | 3 | 1 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 4 | 5 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 1 | 4
  White | 3 | 3 | 3 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: M3541 50 mg + 100 mg + 200 mg + RT: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is classified per the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and defined as any of the following events occurring after first dose of study intervention and judged not to be related to underlying disease or any previous or concomitant medication. Grade (Gr) >=3 non-hematologic toxicity with exception of Nausea, vomiting and diarrhea lasting =<3 days in once per FD; Worsening of preexisting tumor pain associated with tumor lesions for which participant was irradiated in context of this study; Evidence of treatment-related hepatocellular injury for >3 days in the once per FD; Any occurrence of Hy's law; Gr 4 neutropenia lasting for >5 days, Gr 4 thrombocytopenia or Gr 4 anemia that was unexplained by underlying disease; Any toxicity related to study treatment that caused participant to interrupt treatment for not to be able to be treated within 24 hours of the scheduled treatment time.
Time Frame: Baseline up to 5 weeks (including 2 weeks of treatment and 3 weeks of follow-up period)
Population: DLT analysis set included participants who received at least 1 dose of M3541and met at least one of the following criteria: Experienced at least 1 DLT during the DLT evaluation period, regardless of the number of doses of M3541 administered or received at least 80% of planned dose of each treatment, that is, 8 fractions of RT and 8 of 10 M3541 administrations during the treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT
Number analyzed (Participants) | 3 | 4 | 5
Participants | 0 | 0 | 1

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Grade >=3 Adverse Events (AEs), Serious TEAEs and Deaths According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, Version 4.03 (CTCAE V4.03)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are events with start date on or after the date of first dose of study treatment and up to and including 30 days after the last dose of study treatment, or events with start date prior to the date of first dose of study treatment, and worsened in severity or become serious during treatment. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 749 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Participants
  Participants with TEAEs | 3 | 4 | 5 | 3
  Participants with Grade >=3 AEs | 1 | 1 | 1 | 1
  Participants with Serious TEAEs | 0 | 1 | 1 | 0
  Participants with Death | 0 | 4 | 2 | 0

3. Secondary Outcome: Number of Participants With Grade 3 or Higher Laboratory Abnormalities Based on National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Description: The laboratory assessment included measurements hematology and biochemistry parameters. It had been graded according to NCI-CTCAE version 4.03 into Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Life-threatening) and Grade 5 = death. Participants with grade 3 or higher were reported.
Time Frame: Baseline up to Day 44
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Participants
  Hematology | 1 | 1 | 2 | 0
  Biochemistry | 1 | 2 | 3 | 0

4. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Vital signs assessment included blood pressure, pulse rate, body temperature, respiratory rate, and body weight. Notably abnormal vital signs were: Blood pressure: systolic blood pressure >= 140 millimeter of mercury (mmHg) & diastolic blood pressure >=90 mmHg on treatment; Pulse rate >100 beats/min; Body temperature >= 38 degree Celsius (°C) on treatment; Respiratory rate >= 20 breaths/min; Weight (kilogram) > +/-20% from baseline. Number of Participants with abnormalities in vital signs were reported.
Time Frame: Baseline up to 379 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Participants
  Blood Pressure | 1 | 2 | 0 | 0
  Pulse rate | 2 | 2 | 4 | 2
  Body temperature | 0 | 0 | 2 | 0
  Respiratory rate | 1 | 1 | 1 | 1
  Weight | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormalities in Physical Examination Reported as Adverse Events (AEs)
Description: Number of participants with any clinically significant abnormalities in physical examination reported as adverse events with National Cancer Institute Common Terminology Criteria (NCI-CTC) Grade >=3 were presented.
Time Frame: Baseline up to 379 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Participants | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Abnormal Change From Baseline in Electrocardiogram (ECG)
Description: The 12-lead ECG was recorded after the participant was in semi-supine position for at least 5 minutes. The ECG was obtained using a Holter recorder. Number of Participants with abnormal change from baseline in ECG were reported.
Time Frame: Baseline up to 15 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541. Here "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure with normal ECG at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 3 | 0 | 1
Participants |  | 2 |  | 1

7. Secondary Outcome: Number of Participants With Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: BOR was determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). BOR is defined as the best response of any of the complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD is defined as at least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from randomization to 964 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541.
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 2 | 0
  Stable Disease | 1 | 2 | 3 | 3
  Progressive Disease | 1 | 2 | 0 | 0

8. Secondary Outcome: Progression-Free Survival (PFS) Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator
Description: PFS is defined as the time (in months) from first administration of M3541 until the first date of progressive disease (PD) or death due to any cause. PFS was assessed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). PD was defined as at least a 20% increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions. Participants with neither disease progression nor death were censored at the last date of the last tumor assessment that confirmed that their disease had not progressed. Participant wise data reported for this outcome measure.
Time Frame: From first dose of study drug to disease progression or death from any cause, assessed up to 964 days
Population: Safety analysis set included all participants who received at least 1 dose of M3541. The summarized data was not available for this outcome measure, therefore individual data was presented. "Number Analyzed" signifies participants evaluable in respective arm.
Measure: Number; unit: Months
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 3 | 4 | 5 | 3
Months
  Participant-1: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant-1 | 2.92 |  |  |
  Participant-2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant-2 | 11.04 |  |  |
  Participant-3: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant-3 | 1.41 |  |  |
  Participant-4: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant-4 |  | 1.25 |  |
  Participant-5: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant-5 |  | 1.54 |  |
  Participant-6: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant-6 |  | 1.87 |  |
  Participant-7: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant-7 |  | 1.41 |  |
  Participant-8: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant-8 |  |  | 3.55 |
  Participant-9: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant-9 |  |  | 1.97 |
  Participant-10: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant-10 |  |  | 3.55 |
  Participant-11: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant-11 |  |  | 1.84 |
  Participant-12: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant-12 |  |  | 3.15 |
  Participant-13: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant-13 |  |  |  | 2.14
  Participant-14: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant-14 |  |  |  | 1.94
  Participant-15: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant-15 |  |  |  | 1.74

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of M3541
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2.25, 3, 4, 6 hours post-dose on Fraction Day 1; Pre-dose, 2.25 hours post-dose on Fraction Day 2, 5, 6 and 7; Pre-dose, 0.5, 1, 1.5, 2.25, 3, 4, and 6 hours post-dose on Fraction Day 10
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M3541
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of M3541
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of M3541
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Sampling Time Point (AUC[0-last]) of M3541
Description: AUC(0-last) is defined as the area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration. AUC(0-last) will be estimated using the Linear Up Log Down calculation method.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Dose Normalized Area Under the Concentration-Time Curve From Time Zero to the Last Quantifiable Sampling Time Point (AUC[0-last]/Dose) of M3541
Description: The Dose normalized AUC from time zero to the last sampling time (0-last) at which the concentration is at or above the lower limit of quantification. Normalized using the actual dose, using the formula AUC0-last/Dose.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 6 Hour Postdose (AUC[0-6h]) of M3541
Description: Area under the drug concentration-time curve from 0 to 6 hour post dosing for M3541. AUC0-6 was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC[0-inf]) of M3541
Description: AUC0-inf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Dose Normalized Area Under Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC[0-inf]/Dose) of M3541
Description: Dose normalized was calculated as area under the plasma concentration-time curve from time zero to 8 h postdose divided by dose.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Oral Clearance (CL/F) of M3541
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. CL/f = Dose /AUC0-inf. Predicted AUC0-inf should be used.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Oral Clearance at Steady-State (CLss/F) of M3541
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of M3541
Description: The Vz/f was defined as the theoretical volume in which the total amount of required to uniformly distribute to produce the desired plasma concentration. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz/f=Dose/AUC(0-inf)* Lambda(z).
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Apparent Volume of Distribution at Steady-State (Vss/F) of M3541
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss/f after oral dose was influenced by the fraction absorbed.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Accumulation Ratio for Area Under Plasma Concentration-Time Curve From Time Zero to 6 Hour (Racc[AUC0-6]) of M3541
Description: The accumulation ratio to assess the increase in exposure via AUC0-6h. Racc(AUC0-6h)= (AUC0-6h after multiple dose) / (AUC0-6h after single dose).
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Accumulation Ratio for Maximum Observed Plasma Concentration (Racc[Cmax])
Description: The accumulation ratio is to assess the increase in maximum concentration with multiple dosing. Racc(Cmax) = (Cmax after multiple dose)/ (Cmax after single dose).
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of M3541
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of M3541
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Average Plasma Concentration (Cavg) of M3541
Description: Cavg was defined as average plasma concentration.
Time Frame: as for outcome 9
Population: As per changes in planned analysis, the outcome measure related to pharmacokinetic parameters was not assessed.
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Primary Outcome: M3541 300 mg + RT: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: as for outcome 1
Time Frame: Baseline up to 4 weeks (including 2 weeks of treatment and 2 weeks of the follow-up period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M3541 300 mg + RT
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 749 days
Arm/Group | M3541 50 mg + RT | M3541 100 mg + RT | M3541 200 mg + RT | M3541 300 mg + RT
All-Cause Mortality (participants affected / at risk) | 0/3 | 4/4 | 2/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M3541 50 mg + RT (N=3) | M3541 100 mg + RT (N=4) | M3541 200 mg + RT (N=5) | M3541 300 mg + RT (N=3)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M3541 50 mg + RT (N=3) | M3541 100 mg + RT (N=4) | M3541 200 mg + RT (N=5) | M3541 300 mg + RT (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Swelling face (General disorders) | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early per sponsor decision to halt further development of M3541 due to pharmaceutical and PK/pharmacodynamics properties that precluded further clinical development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03225105/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03225105/SAP_001.pdf